CLINICAL TRIAL: NCT06367127
Title: Utility of the Clamping Bean Test (CBT) for Covert Hepatic Encephalopathy Screening in Cirrhotic Patients
Brief Title: Utility of the Clamping Bean Test (CBT) for Covert Hepatic Encephalopathy Screening
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Shanghai Changzheng Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: Pingfanghu
Record Dates: First submitted 2024-01-15; First posted 2024-04-16 (Actual); Last update posted 2024-04-16 (Actual); Status verified 2024-01

CONDITIONS: Hepatic Encephalopathy; Covert Hepatic Encephalopathy
MeSH Terms: conditions — Hepatic Encephalopathy

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Hepatic encephalopathy is a brain dysfunction caused by liver insufficiency and/or porto-systemic shunt. It manifests as a wide spectrum of neurological or psychiatric abnormalities ranging from subclinical alterations to coma. According to the symptoms, it is classified as covert HE (CHE) and overt HE (OHE). CHE can progress to OHE and is associated with reduced driving ability, increased risk of accidents and hospitalization and weakened health-related quality of life, resulting in poor prognosis and socio-economic status. However, due to the absence of readily identifiable clinical symptoms and signs, CHE is often neglected in clinical practice.

Presently, the diagnosis of CHE depends on psychometric and neurophysiological tests, including the psychometric hepatic encephalopathy score (PHES), critical flicker frequency (CFF) test, continuous reaction time (CRT) test, inhibitory control test, the SCAN test, and electroencephalography. Among them, PHES is most widely used and recommended by several guidelines. However, it is difficult to screen CHE among all cirrhotic patients in the clinic using PHES because of the time required and a dependence on trained experts.

Moving beans from one container to another with tweezers involves dexterity, agility and coordination.The hypothesis was that the utility of the Clamping Bean Test (CBT) will enable early screening patients with CHE.

ELIGIBILITY:
Inclusion Criteria:

* written informed consent;
* Age 18-70 years old;
* Patients with clinical diagnosis of liver cirrhosis and without current OHE.

Exclusion Criteria:

* Presence of other uncontrollable neuro-psychiatric or neurological diseases that affect cognitive function, such as Alzheimer's disease, Parkinson's disease, schizophrenia, etc.;
* Clinically diagnosed as overt hepatic encephalopathy(OHE);
* Consumption of hypnotic or sedative drug and psychotropic drug in the past 4 weeks;
* Alcohol consumption >50 g/day within the past 3 months;
* Conditions preventing the patient from completing the test independently (for instance, red-green color blindness, difﬁculty in comprehension).

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Inverstigators will include about 200 healthy volunteers as the healthy control as well. And the data on participants' demographic characteristics, disease history, labratory characteristics and current treatment will be collected.
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2023-10-09 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Number of Beans Clamping in 1 minute | 1 minute
  Moving beans from one container to another with tweezers in one minute, and then count the number of beans

SECONDARY OUTCOMES:
Participants' feedback on CBT1 test | 2 minutes
  Participnants will be asked to complete the questionnaire of the feedback on CBT1 test

CONTACTS AND LOCATIONS:
Overall Officials: Lvping Sun, Study Chair — Shanghai Changzheng Hospital
Locations (1):
- Shanghai Changzheng hospital, Shanghai, China